CLINICAL TRIAL: NCT00645190
Title: A Randomized, Double Blind, Active Control, Flexible Dose, Multicenter Study to Evaluate Galantamine HBr in the Treatment of Alzheimer's Disease:Safety and Effectiveness of an Immediate-release Table Formulation.
Brief Title: A Randomized, Double-blind, Flexible Dose, Multicenter Study to Evaluate the Effectiveness and Safety of Galantamine IR in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005803
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; galantamine
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine HBr

SUMMARY:
The purpose of this randomized, double-blind, active-controlled, flexible dosage, multicenter study is to evaluate the effectiveness and safety of galantamine tablet (16-24mg/day) for 16 weeks in the treatment of mild to moderate Alzheimer's Disease (AD) comparing with Donepezil.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, flexible dosage, multicenter study to evaluate the effectiveness and safety of galantamine tablet in the treatment of mild to moderate AD. The comparator is Donepezil tablet. At least 206 patients were to be randomized in the study. The study consisted of 3 phases: a screening phase, a single-blind run-in phase and a double-blind treatment phase. Screening phase is less than 2 week for eligible assessment; If the patient was taking any anti-dementia drug at screening, he/she had to stop these drugs and enter into the single-blind run-in phase. The patient who did not take any anti-dementia drug can enter into baseline directly. During the single-blind run-in phase, all eligible patients will take placebo twice daily for 4 weeks. Double-blind treatment phase is 16 weeks. At baseline, all patients who are still eligible for inclusion/exclusion criteria will be randomized to either galantamine group or donepezil group at 1:1 ratio, drugs will be taken twice daily by a flexible dose for 16 weeks. Dose will be titrated during the first 9-12 weeks. Dose will be fixed to 16mg/day or 24mg/day based on tolerability of the patient judged by the investigator. The primary effectiveness endpoint is changes in ADAS-cog/11 at week 16 from baseline, secondary endpoint is responder rate in term of ADAS-cog/11. Safety evaluation included adverse events, physical examination, ECG, and safety laboratory tests. Study drug are taken orally twice a day. The treatment duration was 16 weeks. Initial galantamine dose is 8 mg/day, dose was increased to 16mg/day at week 5 and to 24 mg/day at week 9. At week 12, dose was fixed to either 16mg/day or 24mg/day at the discretion of investigators. Initial donepezil dose is 5mg/day, dose was then increased to 10mg/day at week 9. At week 12, dose was fixed to either 5mg/day or 10mg/day at the discretion of investigators.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients diagnosed with mild to moderate probable AD. The diagnosis should have been established in accordance with the classification for probable AD of NINCDS-ADRDA
* MMSE score of 10-24 (inclusive) at screening
* Patients who lived with or had regular daily visits from a responsible caregiver
* .Has signed the informed consent form by subject and assent form by care-giver

Exclusion Criteria:

* Patients with neurodegenerative disorders such as Parkinson's disease
* Patients with some conditions possibly resulting in cognitive impairment, e.g. acute cerebral trauma, infection
* Has evidence of multi-infarct dementia or clinically active cerebrovascular disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2004-03; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Primary endpoint (ADAS-cog/11) decreased 5.4 ± 6.4 and 4 .0 ± 7.3 in galantamine and Donepezil group respectively after 16-week treatment from baseline of 22.5 ± 9.3 and 23.3 ± 9.7 respectively, showing the non-inferiority in term of efficacy.

SECONDARY OUTCOMES:
Secondary endpoint is responder rate. It showed 78% responder rate in galantamine group and 58% responder rate in Donepezil group after 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd. Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

REFERENCES:
- See also: A randomized, active control, double-blind study to evaluate the effectiveness and safety of galantamine for mild to moderate Alzheimer's Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1077&filename=CR005803_CSR.pdf